CLINICAL TRIAL: NCT06954571
Title: A Novel Imaging-Guided Classification System for Completely Endophytic Renal Tumors: Strategies for Optimal Partial Nephrectomy and Clinical Outcome Comparison
Brief Title: Imaging-Guided Classification for Endophytic Renal Tumors: PN Strategies & Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2025K002
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Renal Tumors
Keywords: Renal Tumors
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type1: The tumor is entirely confined within the renal parenchyma, positioned transversely between the ventral and dorsal aspects of the kidney and sagittally within the relatively avascular zone between the upper and lower polar lines, without invading renal pelvis structures.
- Type2: The tumor is located on the ventral aspect of the kidney, adjacent to the anterior wall of the calyx, without involvement of the collecting system . IIb: The tumor is situated on the dorsal aspect of the renal pelvis, closely adjacent to the posterior calyceal wall, without invading the collecting system
- Type3: The tumor occupies the renal hilum region, involves the renal lip or renal sinus, and is closely associated with renal arteries, veins, and the collecting system.

SUMMARY:
Study Title:

Imaging-Guided Classification & Surgical Outcomes in Endophytic Renal Tumors

Study Goal:

This observational study investigates whether an imaging-guided classification system improves partial nephrectomy (PN) outcomes for completely endophytic renal cell carcinoma (RCC).

Main Question:

Does preoperative imaging classification reduce complications (e.g., ischemia time, urinary leakage) in PN for endophytic RCC compared to traditional methods?

Methods:

Patients undergoing PN for endophytic RCC will be grouped based on preoperative imaging classification. Surgical outcomes (complications, renal function) will be tracked for 5 years and compared to non-classified PN cases.

Significance:

Aims to optimize PN planning, minimize risks, and improve long-term renal preservation in complex RCC cases

DETAILED DESCRIPTION:
I. Background of the study Completely endogenous renal cell carcinoma (RCC) is challenging to perform partial nephrectomy (PN) due to the extensive contact area between normal renal parenchyma and RCC and the inability to accurately determine its location from the renal surface.Considering the anatomical complexity and the high risk of complications associated with PN, urologists had favored radical nephrectomy (RN) for completely endophytic RCC to mitigate complications .Advances in robotic-assisted laparoscopic surgery and the use of intraoperative ultrasound have led some clinicians to report prognostic and perioperative outcomes similar to those of RN treatment using PN for these complex endogenous RCCs .Although these studies suggest that PN is an available treatment option for fully endogenous RCC, PN treatment of fully endogenous RCC is usually associated with higher intraoperative and perioperative complications, including longer thermal ischemia time (WIT), higher rates of urinary leakage, and higher rates of positive surgical margins, when compared with PN treatment of non-endogenous RCC .Therefore, performing accurate preoperative planning is essential to help clinicians perform PN for fully endogenous RCC and to minimize associated complications.

In surgery with preservation of renal units, precise preoperative assessment and personalized surgical strategies are crucial for the preservation of postoperative renal function, reduction of complications, and improvement of long-term survival of patients .Therefore, the development of an imaging-based classification system to optimize surgical techniques for completely endophytic tumors is of great clinical importance.

The core objective of this study was to establish a scientific classification system for completely endophytic renal tumors through an imaging-guided preoperative classification method, to explore individualized surgical strategies for preserving renal units, and to analyze their performance in terms of postoperative clinical outcomes to provide new ideas and guidance for clinical practice .

ELIGIBILITY:
Inclusion Criteria:

1. Patients who completed partial resection of completely endogenous renal cancer from January 2018 to November 2024 at the Second Hospital of Tianjin Medical University；
2. Older than 18 years.

Exclusion Criteria:

1. Patients without clinicopathologic, functional or prognosis data；
2. Patients with unilateral multiple renal tumors , solitary kidney , or comorbid severe medical conditions；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who completed partial resection of completely endogenous renal cancer from January 2018 to November 2024 at the Second Hospital of Tianjin Medical University
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Surgical technique | From enrollment to the end of 4 weeks of treatment
  Surgical options for completely endogenous renal cancer include laparoscopic, open, and robotic. The impact on the patient is assessed according to the different surgical modalities.
Trifecta achievement | From enrollment to the end of 4 weeks of treatment
  In renal cancer surgery (particularly partial nephrectomy), the Trifecta achievement consists of:
  * Negative surgical margins (no residual tumor)
  * No perioperative complications (e.g., hemorrhage, urinary leakage)
  * Preservation of renal function (minimal decline in eGFR)
Tumour subtype on histology | From enrollment to the end of 4 weeks of treatment
  The tumor subtypes of renal cancer studied in this study included clear cell carcinoma, papillary carcinoma, and smoky cell carcinoma.
tumor size | From enrollment to the end of 4 weeks of treatment
  It was used to assess the size of the tumor, and in this study, due to the endogenous nature of the tumor, the tumors were generally small, less than 5 cm

SECONDARY OUTCOMES:
age | From enrollment to the end of 4 weeks of treatment
  Patient's age at diagnosis
Gender | From enrollment to the end of 4 weeks of treatment
  Sex of the patient, categorized as male, female.
Tumor side | From enrollment to the end of 4 weeks of treatment
  Split into left and right side.
BMI | From enrollment to the end of 4 weeks of treatment
  Body Mass Index.The formula is: BMI = weight ÷ height squared (weight in kilograms; height in meters)
Smoking history | From enrollment to the end of 4 weeks of treatment
  "0" means current or former smoker, '1' means no smoking. Used to assess whether or not one has smoked. To observe the effect on disease
Alcohol use | From enrollment to the end of 4 weeks of treatment
  "0" indicates current or previous alcohol consumption and '1' indicates no alcohol consumption. Used to assess whether or not one has been drinking. To observe the effect on disease.
Hypertension | From enrollment to the end of 4 weeks of treatment
  "0" means having or currently having high blood pressure and '1' means not having high blood pressure. It is used to assess whether or not a person has ever had a hypertensive disorder.To observe the effect on disease
Diabetes | From enrollment to the end of 4 weeks of treatment
  "0" means current or previous diabetes, '1' means no diabetes. Used to assess for a history of diabetes. To observe the effect on disease
ECOG performance status | From enrollment to the end of 4 weeks of treatment
  0 Fully normal mobility, with no difference in mobility from that before the onset of the disease.
  1. Able to walk freely and engage in light physical activities, including general housework or office work, but unable to engage in heavier physical activities.
  2. Able to walk freely and take care of oneself, but with loss of working ability, and can get up and move around not less than half of the time during the day.
  3. Can only partially take care of oneself, and spends more than half of the day in bed or in a wheelchair.
  4. Bedridden, unable to take care of themselves.
  5. Death Higher scores mean worse.
Charlson comorbidity index | From enrollment to the end of 4 weeks of treatment
  Score 0: Low risk. The patient has no specific co-morbidities included in the CCI score, indicating that the patient is relatively healthy and has a high survival rate.
  Score 1-2: Moderate risk. Patients may have one or two milder co-morbidities, but overall risk is relatively low.
  Score 3-4: Moderate to high risk. Patients may have a moderate burden of co-morbidities and may have reduced survival.
  Score 5-6: High risk. Patients have a high burden of co-morbidities and may require closer monitoring and care.
  Score 7 and above: Very high risk. The patient has a more severe burden of co-morbidities and may have significantly reduced survival and a higher risk of treatment.
ASA score | From enrollment to the end of 4 weeks of treatment
  1. Physical health, good development and nutrition, normal function of organs. Perioperative mortality rate 0.06%-0.08%;
  2. Mild coexisting diseases other than surgical diseases, with sound functional compensation. Perioperative mortality rate 0.27%-0.40%;
  3. Severe coexisting conditions with limited physical activity, but still able to cope with daily activities. Perioperative mortality rate 1.82%-4.30%;
  4. Severe coexisting conditions with loss of ability to perform daily activities and frequent life threatening situations. Perioperative mortality rate 7.80%-23.0%;
  5. Dying patients who have difficulty sustaining life for 24 hours regardless of surgery. Perioperative mortality rate 9.40%-50.7%;
  6. Confirmed brain death with organs intended for organ transplantation.
P.A.D.U.A. score | From enrollment to the end of 4 weeks of treatment
  The scores are 0, 1, 2, 3 and 4, ranging from "none" to "very serious", respectively.
R.E.N.A.L. score | From enrollment to the end of 4 weeks of treatment
  The R.E.N.A.L. scoring system is based on the anatomical features of renal tumors, including tumor size (R), convexity (E), relationship to the renal sinus and collecting system (N), ventral or dorsal renal location (A), location along the longitudinal axis of the kidney (L), and relationship to the renal hilum (h), and quantitatively evaluates each aspect based on the scores.
  Higher scores mean worse.
operative time | From enrollment to the end of 4 weeks of treatment
  The time it takes the doctor to make the cut and the time it takes to close the incision.
estimated blood loss | From enrollment to the end of 4 weeks of treatment
  By intraoperative blood loss, we actually mean loss of circulating blood volume
warm ischemia time | From enrollment to the end of 4 weeks of treatment
  The length of time between blocking the blood supply to the kidneys, the state of persistent ischemia at room temperature, and the restoration of the blood supply.
Postoperative length of hospital stay | From enrollment to the end of 8 weeks of treatment
  Length of hospitalization of patients after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Wang K, Zhang J, Zhou W, Liu Y, Yao Z, Yao J, Liu Y, Zhang J, Liu K, Li G. A Novel Imaging-Guided Classification System for Completely Endophytic Renal Tumors: Strategies for Optimal Partial Nephrectomy and Clinical Outcome Comparison. Ann Surg Oncol. 2025 Nov 22. doi: 10.1245/s10434-025-18756-x. Online ahead of print. PMID 41273672